CLINICAL TRIAL: NCT00987675
Title: An Evaluation of Lesion Control Using Focal Ablation With High Intensity Focused Ultrasound in the Treatment of Non-Metastatic Progressive Prostate Cancer
Brief Title: High-Intensity Focused Ultrasound Ablation in Treating Patients With Progressive Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000650138; UCLH-09-H0714-7
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Intensity Focused Ultrasound Ablation

INTERVENTIONS:
Other: pharmacological study
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: high-intensity focused ultrasound ablation
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: High-intensity focused ultrasound ablation uses high-energy sound waves to kill tumor cells.

PURPOSE: This phase II trial is studying the side effects of high-intensity focused ultrasound ablation and to see how well it works in treating patients with progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the side effects and patient-reported quality of life outcomes of the index (largest) lesion treatment with high-intensity focused ultrasound ablation in patients with progressive ≤ T3b, N0, M0 prostate cancer.

Secondary

* To determine the success of this treatment by demonstrating the absence of cancer in the treated or ablated area on the 6 month post-treatment transrectal ultrasound biopsy.
* To evaluate the prostate-specific antigen (PSA) kinetics after index lesion ablation treatment in these patients.
* To evaluate the proportion of these patients who, after undergoing index lesion control treatment, require androgen blockade at the 12-month follow-up.

OUTLINE: Patients undergo transrectal high-intensity focused ultrasound ablation (HIFU) to the index lesion and other identifiable secondary lesions. Patients are evaluated at 6 months and may repeat HIFU treatment.

Patients undergo MRI and ultrasound at baseline and periodically thereafter, and blood samples are collected periodically for PSA, renal function, full blood count, and testosterone levels. Patients also complete questionnaires (IPSS, IPSS-QOL, ICS, FACT-P, and IIEF-5) at baseline; at 6 weeks; and at 3, 6, 9 and 12 months.

After completion of study treatment, patients are followed at 2 and 6 weeks and at 3, 6, 9, and 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer on transrectal ultrasound or transperineal template prostate biopsies meeting the following criteria:

  * Stage ≤ T3b, N0, M0 disease
  * Gleason score ≤ 8
  * Serum PSA ≤ 20 ng/mL
  * No metastatic disease and nodal spread by staging CT or MRI

    * Negative bone scan within the past 6 months
* Index lesion or other secondary lesions with a volume of ≥ 0.5 cc by MRI

  * Secondary lesions are included in the treatment provided ≥ 1 neurovascular bundle and 40-50% of prostatic tissue can be preserved

PATIENT CHARACTERISTICS:

* Able to tolerate a transrectal ultrasound
* Able to undergo major surgery as assessed by a consultant anesthesiologist
* Able to undergo MRI scanning (i.e., no severe claustrophobia, permanent cardiac pacemaker, metallic implant)
* No urethral stricture or presence of metal implants or stents in the urethra
* No prostatic calcification or cysts (on transrectal ultrasound) that would interfere with effective delivery of HIFU therapy
* No allergy to latex

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy
* No prior treatment with any of the following:

  * Transurethral resection of the prostate or equivalent procedures within the past 2 years
  * High-intensity focused ultrasound ablation (HIFU)
  * Cryosurgery
  * Thermal or microwave therapy to the prostate
* No prior significant rectal surgery that prevents insertion of the transrectal HIFU probe
* More than 12 months since prior androgen suppression or hormone treatment for prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Side effects and patient-reported quality of life after treatment as measured by IPSS, IPSS-QOL, ICS, FACT-P, and IIEF-5 questionnaires at baseline, 6 weeks, and 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Success of treatment as demonstrated by the absence of cancer at 6 months
PSA kinetics after completion of treatment
Proportion of patients requiring androgen blockade at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Uddinn Ahmed, MD — University College London Hospitals
Locations (1):
- University College Hospital, London, England, United Kingdom